CLINICAL TRIAL: NCT03227250
Title: Effects of Bilateral Pallidal Deep Brain Stimulation on Freezing of Gait in Parkinson's Diseases
Brief Title: Effects of Bilateral GPI DBS on Freezing of Gait in PD
Acronym: PD GPI DBS
Status: Completed | Type: Observational
Sponsor: Haiyan Zhou (Other)
Responsible Party: Sponsor-Investigator, Haiyan Zhou, attending neurologist, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: GPIFOG
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: freezing of gait; Parkinson disease; GPi
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GPI DBS: patients who had freezing of gait and underwent deep brain stimulation (DBS) of the globus pallidus interna (GPi)

SUMMARY:
This study aims to evaluate the effect of deep brain stimulation in the the globus pallidus (Gpi) on freezing of gait in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion criteria: (1) idiopathic PD, according to the MDS Parkinson's Disease Society Diagnostic Criteria17; (2) bilateral GPi-DBS implant according to a careful consideration of patients' symptom profiles (e.g., existence and severity of dyskinesia, dystonia, axial symptoms, or cognitive and mood problems); (3) onset of PD at or before 70 years of age; and (4) disease duration of more than 3 years at the time of surgery.

Patients were excluded if they had unstable vital signs or medical and psychiatric comorbidities at the time of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who underwent GPI DBS.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Changs in the score of Timed Up and Go Test | baseline, 12 month

SECONDARY OUTCOMES:
Change of the score in GFQ | baseline, 12 month
Change of the score in FoG total time of TUG test | baseline, 12 month
Change of the score in FoG Episodes of TUG test | baseline, 12 month
Change of the score in Proportion of FoG of TUG test | baseline, 12 month
Change of the score in Longest FoG duration of TUG test | baseline, 12 month

OTHER OUTCOMES:
Change of the scores in MDS-UPDRS | baseline, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Zhou, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Shengdi Chen, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Dianyou Li, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Bomin Sun, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Wei Hu, Principal Investigator — University of Florida
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No